CLINICAL TRIAL: NCT00216892
Title: Different Treatment Regimens of Calcipotriol Cream and Combination (Calcipotriol/Betamethasone Dipropionate) Ointment in Psoriasis Vulgaris
Brief Title: Efficacy and Safety of Calcipotriol Cream and (Calcipotriol + Betamethasone Dipropionate) Ointment in Psoriasis Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCB 0402 INT
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; Betamethasone

INTERVENTIONS:
Drug: Calcipotriol, (calcipotriol + betamethasone)

SUMMARY:
Patients with psoriasis vulgaris of the trunk and/or limbs are randomised to treatment with:

1. 4 weeks of ointment containing calcipotriol and betamethasone dipropionate followed by 8 weeks of calcipotriol cream
2. 4 weeks of (calcipotriol plus betamethasone dipropionate) ointment followed by 8 weeks of calcipotriol cream on weekdays/ (calcipotriol plus betamethasone dipropionate) ointment on weekends
3. 4 weeks of (calcipotriol plus betamethasone dipropionate) ointment followed by 8 weeks of vehicle of calcipotriol cream

The objective is to compare the efficacy and safety of the different treatment regimens

DETAILED DESCRIPTION:
A phase IV study of different treatment regimens of calcipotriol 50 mcg/g cream and combination (calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate)) ointment following treatment with combination ointment in psoriasis vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis vulgaris of trunk and/or limbs

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1032
Dates: Start 2005-04; Study Completion 2005-12

PRIMARY OUTCOMES:
Efficacy of regimen (a) versus regimen (c) by % change in PASI at week 12

SECONDARY OUTCOMES:
Efficacy of regimen (b) versus regimen (c) at week 12, safety of regimen (a) versus (c), safety of regimen (b) versus (c)

CONTACTS AND LOCATIONS:
Overall Officials: S White, MD, Principal Investigator — Clatterbridge Hospital, Department of Dermatology
Locations (7):
- Universitair Ziekenhuis, Ghent, Belgium
- Dermatrials Research Dermatology Centre, Hamilton, Ontario, Canada
- Hôpital Nord, Service de Dermatologie, Saint-Etienne, France
- Klinikum der Goethe-Universität, Zentrum für Dermatologie und Venerologie, Frankfurt, Germany
- Canisius-Wilhelmina Ziekenhuis, Nijmegen, Netherlands
- Hospital Mutua de Terrassa Dermatology Service, Terrassa, Spain
- Clatterbridge Hospital, Department of Dermatology, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en